CLINICAL TRIAL: NCT05249543
Title: Transdiagnostic Versus Diagnosis-specific Cognitive-behavioral Therapy for Anxiety Disorders: a Randomized Controlled Pilot Study
Brief Title: Transdiagnostic Versus Diagnosis-specific Cognitive-behavioral Therapy
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Benjamin Bohman, Study Principal Investigator, Karolinska Institutet
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: KI-2021-05587-01
Record Dates: First submitted 2022-01-14; First posted 2022-02-21 (Actual); Last update posted 2025-03-04 (Actual); Status verified 2025-03

CONDITIONS: Panic Disorder; Generalized Anxiety Disorder; Social Anxiety Disorder; Obsessive-Compulsive Disorder; Posttraumatic Stress Disorder
Keywords: Transdiagnostic Treatment; Unified Protocol; Cognitive-Behavioral Therapy; Anxiety Disorders; Pilot Study
MeSH Terms: conditions — Panic Disorder; Generalized Anxiety Disorder; Phobia, Social; Obsessive-Compulsive Disorder; Stress Disorders, Post-Traumatic; Anxiety Disorders

STUDY DESIGN:
Intervention Model Description: Participants are consecutively included in the study and randomly allocated to treatment condition using a 1:1 ratio.
Who Masked: Investigator, Outcomes Assessor
Masking Description: Investigators are blinded to treatment condition in the analysis phase. Outcome assessors conducting diagnostic interviews and clinical severity ratings are blinded to treatment condition at post assessment.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Unified protocol (Experimental): Transdiagnostic cognitive-behavioral therapy focusing on emotional processes central to the development and maintenance of anxiety disorders, particularly neuroticism.
  Interventions: Behavioral: Unified protocol
- Diagnosis-specific cognitive-behavioral therapy (Active Comparator): Cognitive-behavioral therapy specifically designed for a particular anxiety disorder as specified in evidence-based treatment protocols, which are commonly based on a specific theory or model of the development and maintenance of an anxiety disorder.
  Interventions: Behavioral: Diagnosis-specific cognitive-behavioral therapy

INTERVENTIONS:
Behavioral: Unified protocol — Transdiagnostic cognitive-behavioral therapy
  Arms: Unified protocol
Behavioral: Diagnosis-specific cognitive-behavioral therapy — Diagnosis-specific cognitive-behavioral therapy
  Arms: Diagnosis-specific cognitive-behavioral therapy

SUMMARY:
The primary aim of the pilot study is to investigate the feasibility of conducting a randomized controlled trial (RCT) comparing the effects of transdiagnostic and diagnosis-specific cognitive-behavioral therapy (CBT) for patients with anxiety disorders in routine psychiatric outpatient care in Stockholm, Sweden. It is hypothesized that an RCT is feasible in terms of recruitment, retention, therapist competence and adherence to treatments, and that the treatments are well received by participants.

DETAILED DESCRIPTION:
Aim

The primary aim of the pilot study is to investigate the feasibility of conducting an RCT comparing the the effects of two types of protocol-based individual CBT for patients with anxiety disorders: transdiagnostic CBT using the unified protocol (UP) and diagnosis-specific CBT using single disorder protocols (SDP). The aim of a future RCT is to replicate the only equivalence RCT of the UP and SDPs for patients with anxiety disorders (Barlow et al., 2017). Feasibility is investigated in terms of a) recruitment of participants across diagnoses, b) retention of participants and data loss at post treatment, c) therapist competence in and adherence to the UP and SDPs, d) treatment credibility and expectancy of improvement and treatment satisfaction, and e) adverse effects. A secondary aim is to explore the effects of the treatments in terms of a) clinical severity of diagnosis, b) anxiety and depressive symptoms, and c) functional impairment and quality of life.

Design

Randomized controlled design by which the UP is compared to SDPs. Randomization of participants is conduced using a 1:1 ratio. A sequence of random numbers are generated per therapist by an independent assistant using an online random number service. The study is conducted in routine psychiatric outpatient care at clinics in Stockholm, Sweden.

Participants

For inclusion and exclusion criteria, see other data elements. To investigate the feasibility of an RCT and expecting a dropout rate of 20% consistent with prior research of CBT for anxiety disorders, we believe that 76 participants is an appropriate number. In addition, prior to recruitment of participants for treatment, 16 participants (four per therapist) are recruited for assessment of therapist competence and adherence to the UP and SDPs. Therapists are psychologists with training in SDPs. As their competence and adherence are assessed, therapists are also participants in the study.

Assessment

Diagnostic assessment is conducted using the Mini International Neuropsychiatric Interview (Sheehan et al., 1998). Clinical severity of diagnosis is assessed using the Clinical Severity Rating (CSR; Brown & Barlow, 2014), which is rated 0-8 with 4 and above indicating meeting a diagnosis. For feasibility and treatment effects measures, see other data elements.

Feasibility measures

Participant recruitment. We expect to be able to recruit at least seven participants per month with four therapists.

Attrition. A common attrition rate in studies of CBT for anxiety disorders is 20%. I the 2017 equivalence RCT by Barlow and colleagues, 88% of participants in the UP condition and 69% of participants in the SDP condition completed treatment (defined as attending at least 75% of sessions). Thus, we expect an attrition rate of 20% at the most in respective treatment condition.

Competence in and adherence to the UP and SDPs. Prior to participant recruitment, therapists record treatment sessions on audio with participants who are not treated in the study and these audio-recordings are coded by independent raters to assess therapist competence and adherence to the UP and SDPs. Assessment of competence in and adherence to the UP is conducted using the UP Adherence and Competence Scale (Boswell et al., 2013). This assessment is included in the UP training of therapists and is conducted for all treatment modules used with one participant exclusively recruited for training purposes. Assessment of competence in diagnosis-specific CBT is conducted using the Cognitive Therapy Scale-Revised (Blackburn et al., 2001), and adherence using the Adherence to Cognitive-Behavioral Therapy Scale (Bergvall & Bohman, 2018). For diagnosis-specific CBT, estimates of competence and adherence are based on three treatment sessions with three different participants per therapist recorded on audio and coded by independent raters. These three participants are not treated in the study. As for participants treated in the study, participants who are recruited only for training and assessment purposes provide written informed consent to take part in the study.

Perceptions of the UP and SDPs and study procedures. Both patients and therapists respond to surveys exploring the provision or receipt of the treatments. Patients also respond to questions covering study procedures, including the assessment procedure and number of measures at different assessment points.

Treatment credibility and expectancy of improvement is assessed at session 2 using the Credibility/Expectancy Questionnaire (Devilly & Borkovec, 2000). Treatment satisfaction is assessed at post treatment using the Client Satisfaction Questionnaire (Attkison & Greenfield, 1996). Adverse effects are assessed during treatment by therapists reporting on suicidal or other negative events, and by using the Negative Effects Questionnaire (Rozental et al., 2019) or a similar measure at post assessment.

Treatment effects measures

A preliminary exploration of treatment effects and assessment of a purported mediator are conducted. Primary treatment effects measure is clinical severity of diagnosis assessed using the CSR. The CSR is used at pre treatment by the therapist conducting the assessment, and at post treatment by an independent therapist who is blind to treatment condition.

In addition, treatment effects are explored in both conditions using self-report measures. General symptoms of anxiety and depression are assessed at pre and post treatment, and at each session using the Overall Anxiety Severity and Impairment Scale (OASIS; Norman et al., 2006) and the Overall Depression Severity and Impairment Scale (ODSIS; Bentley et al., 2014), respectively. These measures are used as part of the UP, and are also administered to participants in the SDP condition.

The following diagnosis-specific self-report measures, corresponding to the principal diagnosis, are responded to at pre and post treatment: the Panic Disorder Severity Scale-Self-Rated (Houck et al., 2002) for panic disorder, the Obsessive Compulsive Inventory-Revised (Foa et al., 2002) for obsessive-compulsive disorder, the Penn State Worry Questionnaire (Meyer et al., 1990) for generalized anxiety disorder, the Liebowitz Social Anxiety Scale-Self-Report (Fresco et al., 2001) for social anxiety, and the Posttraumatic Stress Disorder Checklist-5 (Blevins et al., 2015) for post-traumatic stress disorder.

At pre and post treatment, functional impairment is assessed using the World Health Organization Disability Assessment Schedule (World Health Organization, 2010), and quality of life using the EuroQol Five Dimensional Questionnaire (EuroQol Group, 1990). In addition, neuroticism, the purported mediator of the UP (Barlow et al., 2017; Sauer-Zavala et al., 2020) is assessed at pre and post treatment and at each session using the neuroticism subscale of the Eysenck Personality Questionnaire Revised - Short Form (Eysenck et al., 1985). The purpose of assessing neuroticism is to investigate adherence to multiple assessments, and to evaluate sensitivity to change.

Treatments

The UP is implemented using the Swedish translation of the published protocol (Barlow et al., 2018a, 2018b), and SDPs using evidence-based protocols recommended in clinical guidelines (e.g., prolonged exposure for post-traumatic stress disorder; Foa et al., 2007). All treatments consist of 12-18 sessions, and the number of sessions per diagnosis are matched for the UP and SDPs, so the treatment dose is the same across treatment conditions.

Procedure

Therapists receive training in the UP. Each therapist provides both the UP and SDPs in equal amounts. During treatment, therapists receive supervision in both conditions. Eligible patients are provided with oral and written study information and are invited to participate by the therapist who conduct assessment, including a diagnostic interview. Patients who consent to participate respond to self-report measures and are randomly allocated to receive the UP or an SDP. Following the last session, a diagnostic interview is conducted by an independent therapist blind to treatment condition, and participants respond to the same self-report measures.

Data analysis

Feasibility measures are analyzed primarily using descriptive statistics. Preliminary treatment effects measures are analyzed according to the intention-to-treat principle using multilevel modeling. Model-based effect sizes with 95% confidence intervals are calculated using equations suggested in Feingold (2015). In addition, based on Jacobson and Truax (1991), reliable change and clinical significance are calculated.

References

Attkison, C. C., & Greenfield, T.K. . (1996). The client satisfaction questionnaire (CSQ) scales and the service satisfaction Scale-30 (SSS-30). In L. I. D. Sederer, B. (Ed.), Outcomes assessment in clinical practice. (pp. 120-127). Williams & Wilkins.

Barlow, D. H., Farchione, T. J., Bullis, J. R., Gallagher, M. W., Murray-Latin, H., Sauer- Zavala, S., Bentley, K. H., Thompson-Hollands, J., Conklin, L. R., Boswell, J. F., Ametaj, A., Carl, J. R., Boettcher, H. T., & Cassiello-Robbins, C. (2017). The Unified Protocol for Transdiagnostic Treatment of Emotional Disorders compared with diagnosis-specific protocols for anxiety disorders: a randomized clinical trial. JAMA Psychiatry, 74(9), 875-884.

Barlow, D. H., Sauer-Zavala, S., Farchione, T. J., Murray Latin, H., Ellard, K. K., Bullis, J. R., Bentley, K. H., Boettcher, H. T., & Cassiello-Robbins, C. (2018a). Unified protocol for transdiagnostic treatment of emotional disorders: workbook (2nd ed.). Oxford University Press.

Barlow, D. H., Farchione, T. J., Sauer-Zavala, S., Murray Latin, H., Ellard, K. K., Bullis, J. R., Bentley, K. H., Boettcher, H. T., & Cassiello-Robbins, C. (2018b). Unified protocol for transdiagnostic treatment of emotional disorders: therapist guide (2nd ed.). Oxford University Press.

Bentley, K. H., Gallagher, M. W., Carl, J. R., & Barlow, D. H. (2014). Development and validation of the Overall Depression Severity and Impairment Scale. Psychol Assess, 26(3), 815-830.

Bergvall, H., & Bohman, B. (2018). The Adherence to Cognitive-Behavioral Therapy Scale: Observer Version. Unpublished.

Blackburn, I.-M., James, I. A., Milne, D. L., Baker, C., Standart, S., Garland, A., & Reichelt, F. K. (2001). The Revised Cognitive Therapy Scale (CTS-R): psychometric properties. Behav Cogn Psychother, 29, 431-446.

Blevins, C. A., Weathers, F. W., Davis, M. T., Witte, T. K., & Domino, J. L. (2015). The Posttraumatic Stress Disorder Checklist for DSM-5 (PCL-5): Development and Initial Psychometric Evaluation. J Trauma Stress, 28(6), 489-498.

Boswell, J. F., Gallagher, M. W., Sauer-Zavala, S. E., Bullis, J., Gorman, J. M., Shear, M. K., Woods, S., & Barlow, D. H. (2013). Patient characteristics and variability in adherence and competence in cognitive-behavioral therapy for panic disorder. J Consult Clin Psychol, 81(3), 443-454.

Brown, T. A., & Barlow, D. H. (2014). Anxiety and Related Disorders Interview Schedule for DSM-5-Lifetime Version. Oxford University Press.

Devilly, G. J., & Borkovec, T. D. (2000). Psychometric properties of the credibility/expectancy questionnaire. J Behav Ther Exp Psychiatry, 31(2), 73-86.

Eysenck, S. B., Eysenck, H. J., & Barrett, P. (1985). A revised version of the psychoticism scale. Personality and Individual Differences, 6, 21-29.

EuroQol Group. (1990). EuroQol - a new facility for the measurement of health-related quality of life. Health Policy, 16(3), 199-208.

Feingold, A. (2015). Confidence interval estimation for standardized effect sizes in multilevel and latent growth modeling. J Consult Clin Psychol, 83(1), 157-168.

Foa, E. B., Hembree, E. A., & Rothbaum, B. O. (2007). Prolonged exposure therapy for PTSD: emotional processing of traumatic experiences. Oxford University Press.

Foa, E. B., Huppert, J. D., Leiberg, S., Langner, R., Kichic, R., Hajcak, G., & Salkovskis, P. M. (2002). The Obsessive-Compulsive Inventory: development and validation of a short version. Psychol Assess, 14(4), 485-496.

Fresco, D. M., Coles, M. E., Heimberg, R. G., Liebowitz, M. R., Hami, S., Stein, M. B., & Goetz, D. (2001). The Liebowitz Social Anxiety Scale: a comparison of the psychometric properties of self-report and clinician-administered formats. Psychol Med, 31(6), 1025-1035.

Houck, P. R., Spiegel, D. A., Shear, M. K., & Rucci, P. (2002). Reliability of the self-report version of the Panic Disorder Severity Scale. Depress Anxiety, 15(4), 183-185.

Jacobson, N. S., & Truax, P. (1991). Clinical significance: a statistical approach to defining meaningful change in psychotherapy research. J Consult Clin Psychol, 59(1), 12-19.

Meyer, T. J., Miller, M. L., Metzger, R. L., & Borkovec, T. D. (1990). Development and validation of the Penn State Worry Questionnaire. Behav Res Ther, 28(6), 487-495.

Norman, S. B., Cissell, S. H., Means-Christensen, A. J., & Stein, M. B. (2006). Development and validation of an Overall Anxiety Severity And Impairment Scale (OASIS). Depress Anxiety, 23(4), 245-249.

Rozental, A., Kottorp, A., Forsstrom, D., Mansson, K., Boettcher, J., Andersson, G., Furmark, T., & Carlbring, P. (2019). The Negative Effects Questionnaire: psychometric properties of an instrument for assessing negative effects in psychological treatments. Behav Cogn Psychother, 47(5), 559-572.

Sauer-Zavala, S., Fournier, J. C., Jarvi Steele, S., Woods, B. K., Wang, M., Farchione, T. J., & Barlow, D. H. (2020). Does the unified protocol really change neuroticism? Results from a randomized trial. Psychol Med, 1-10.

Sheehan, D. V., Lecrubier, Y., Sheehan, K. H., Amorim, P., Janavs, J., Weiller, E., Hergueta, T., Baker, R., & Dunbar, G. C. (1998). The Mini-International Neuropsychiatric Interview (M.I.N.I.): the development and validation of a structured diagnostic psychiatric interview for DSM-IV and ICD-10. J Clin Psychiatry, 59 Suppl 20, 22- 33;quiz 34-57.

World Health Organization. (2010). Measuring Health and Disability: Manual for WHO Disability Assessment Schedule WHODAS 2.0. WHO.

ELIGIBILITY:
Inclusion Criteria:

* 18-65 years of age,
* Being able to speak Swedish without interpreter support,
* A principal diagnosis of panic disorder, generalized anxiety disorder, social anxiety disorder, obsessive-compulsive disorder, or posttraumatic stress disorder, and
* Pharmacological treatment (if any) that is stable six weeks prior to treatment start

Exclusion Criteria:

* Current diagnosis of psychotic disorder, bipolar disorder, or moderate to severe substance use disorder,
* Moderate to severe risk of suicide,
* Psychiatric, somatic, or social problems which require other management or intervention than cognitive-behavioral therapy, and
* Other simultaneous psychological treatment

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-representation of gender identity: female, male, other.
Enrollment: 76 (Estimated)
Dates: Start 2022-03-01 (Actual); Primary Completion 2025-09 (Estimated); Study Completion 2025-09 (Estimated)

PRIMARY OUTCOMES:
Feasibility measure 1 | Prior to pre assessment, up to 1 month
  Recruitment of participants: the number of participants per diagnosis included in the study
Feasibility measure 2 | During treatment, up to 18 weeks
  Attrition: the number of participants dropping out of treatment
Feasibility measure 3 | Prior to pre assessment, up to 6 months
  Therapist competence in and adherence to the unified protocol according to the UP Adherence and Competence Scale, and diagnosis-specific cognitive-behavioral therapy according to the Cognitive Therapy Scale-Revised
Feasibility measure 4 | During treatment Week 2
  Treatment credibility and expectancy of improvement according to the Credibility/Expectancy Questionnaire
Feasibility measure 5 | At post assessment, up to 18 weeks
  Treatment satisfaction according to the Client Satisfaction Questionnaire
Feasibility measure 6 | At post assessment, up to 18 weeks
  Adverse effects according to the Negative Effects Questionnaire

SECONDARY OUTCOMES:
Change in Clinical Severity Rating - primary outcome measure for preliminary exploration of treatment effects | Change from baseline at up to 18 weeks
  Diagnoses are assigned a dimensional clinical severity rating on a scale from 0 (no symptoms) to 8 (extremely severe symptoms), with a rating of 4 or higher (definitely disturbing or disabling) representing the clinical threshold for diagnostic criteria. Observer-assessed.
Change in Overall Anxiety Severity and Impairment Scale | Change from baseline at up to 18 weeks
  Self-reported general anxiety
Change in Overall Depression Severity and Impairment Scale | Change from baseline at up to 18 weeks
  Self-reported depression
Change in Diagnosis-specific symptoms measures | Change from baseline at up to 18 weeks
  Self-reported panic symptoms, generalized anxiety symptoms, social anxiety symptoms, obsessive-compulsive symptoms, and posttraumatic stress symptoms, respectively.
Change in World Health Organization Disability Assessment Schedule | Change from baseline at up to 18 weeks
  Self-reported functional impairment
Change in EuroQol Five Dimensional Questionnaire | Change from baseline at up to 18 weeks
  Self-reported quality of life
Change in Eysenck Personality Questionnaire - Revised | Change from baseline at up to 18 weeks
  Neuroticism subscale, a measure of the purported mediator of the unified protocol

CONTACTS AND LOCATIONS:
Overall Officials: Benjamin Bohman, PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- WeMind, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No